CLINICAL TRIAL: NCT05538754
Title: Post-Market Evaluation of the EVO ICL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Staar Surgical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP22-01
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Myopia; Myopic Astigmatism
Keywords: nearsightedness; phakic IOL; toric ICL; ICL; TICL; EVO; astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will undergo phakic eye surgery to have the STAAR EVO Implantable Collamer Lens (ICL) implanted in one or both eligible eyes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EVO ICL (Other): STAAR EVO implantable collamer lens (ICL) for the correction or reduction of myopia or myopia with astigmatism.
  Interventions: Device: EVO ICL

INTERVENTIONS:
Device: EVO ICL — The EVO ICL is intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior capsule of the human crystalline lens.

SUMMARY:
The objective of this study is to assess the rate of early intraocular pressure (IOP) increases following implantation of EVO/EVO+ Implantable Collamer Lens (ICL).

DETAILED DESCRIPTION:
This study will be conducted at up to 10 sites in the US, by surgeons qualified by experience and training to implant the EVO/EVO+ lens.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to high myopia correctable with available EVO ICL powers.
* Moderate to high myopic with astigmatism correctable with available EVO ICL powers.
* Stable refractive history within 0.50 D cylinder for 1 year prior to implantation.
* Stable refractive history within 0.50 D for spherical equivalent 1 year prior to implantation.
* Able and willing to return for scheduled follow-up examinations after surgery.
* Able to read, understand and provide written informed consent on the Institutional Review Board (IRB) approved informed consent form (ICF) and provide authorization as appropriate for local privacy regulations.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Ocular hypertension or glaucoma.
* Insulin dependent diabetes or diabetic retinopathy.
* History of previous ocular surgery.
* Monocular.
* Pregnant or nursing women, or those who plan to become pregnant over the course of this clinical study or has another condition with associated fluctuation of hormones that could lead to refractive changes.
* Other protocol-specified exclusion criteria may apply.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Egamino, PhD, Study Director — Staar Surgical Company
Locations (8):
- United States (8):
  - Aloha Laser Vision, LLC, Honolulu, Hawaii
  - Durrie Vision, Overland Park, Kansas
  - Kugler Vision, PC, Omaha, Nebraska
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Key-Whitman Eye Center, Dallas, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 205 subjects were enrolled and treated at 8 clinical sites in the United States. The first enrolled subject underwent surgery in the primary eye on 05 Oct 2022 and the last eye was implanted on 21 Sep 2023.
Units Other Than Participants: Eyes
Groups:
- Primary Eyes: First implanted eyes of enrolled subjects. EVO/EVO+ICL: The investigational lenses are intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior capsule of the human crystalline lens.
- Fellow Eyes: Second implanted eyes of enrolled subjects. EVO/EVO+ICL: The investigational lenses are intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior capsule of the human crystalline lens.
Period: Overall Study
Arm/Group | Primary Eyes | Fellow Eyes
Started | 205; 205 Eyes | 205; 203 Eyes
Completed | 205; 205 Eyes | 205; 203 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: Baseline data were collected on the whole participant level
Groups:
- EVO ICL: Enrolled patients who underwent surgery with an ICL lens in at least one eye.
Arm/Group | EVO ICL
Number analyzed (Participants) | 205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 205
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126
  Male | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33
  Not Hispanic or Latino | 172
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 176
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 205

OUTCOME MEASURES:

1. Primary Outcome: Elevated Intraocular Pressure (IOP) in Primary Eyes ≥ 30 mmHg
Description: The number of primary (first implanted) eyes that have elevated intraocular pressure measuring ≥ 30 mmHg as assessed with applanation tonometry which is a noninvasive test that measures the pressure inside the eye by flattening a part of the cornea.
Time Frame: 1-6 hours postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Primary Eyes: First implanted eyes of enrolled patients. EVO/EVO+ICL: The investigational lenses are intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior capsule of the human crystalline lens.
Arm/Group | Primary Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 205
Eyes | 15

2. Primary Outcome: Elevated Intraocular Pressure (IOP) in Primary Eyes ≥ 40 mmHG
Description: The number of primary (first implanted) eyes that have elevated intraocular pressure measuring ≥ 40 mmHG as assessed with applanation tonometry which is a noninvasive test that measures the pressure inside the eye by flattening a part of the cornea.
Time Frame: 1-6 hours postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Primary Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 205
Eyes | 4

3. Secondary Outcome: Elevated Intraocular Pressure (IOP) in Fellow Eyes ≥ 30 mmHg
Description: The number of fellow (second implanted) eyes that have elevated intraocular pressure measuring ≥ 30 mmHg as assessed with applanation tonometry which is a noninvasive test that measures the pressure inside the eye by flattening a part of the cornea.
Time Frame: 1-6 hours postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Fellow Eyes: Second implanted eyes of enrolled patients. EVO/EVO+ICL: The investigational lenses are intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior capsule of the human crystalline lens.
Arm/Group | Fellow Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 203
Eyes | 16

4. Secondary Outcome: Elevated Intraocular Pressure (IOP) in Fellow Eyes ≥ 40 mmHG
Description: The number of fellow (second implanted) eyes that have elevated intraocular pressure measuring ≥ 40 mmHG as assessed with applanation tonometry which is a noninvasive test that measures the pressure inside the eye by flattening a part of the cornea.
Time Frame: 1-6 hours postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Fellow Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 203
Eyes | 6

5. Other Pre Specified Outcome: Cumulative Rates of Increased Intraocular Pressure (IOP) in All Eyes Attributed to Retained OVD
Description: Rates of elevated intraocular pressure in all (primary + fellow) eyes attributed to retained Ophthalmic Viscoelastic Device (OVD) a clear gel-like material used in eye surgery to maintain the volume and shape of the anterior chamber of the eye.
Time Frame: 1-6 hours postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- All Treated Eyes: EVO/EVO+ ICL: the investigational lenses are intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior chamber of the human crystalline lens.
Arm/Group | All Treated Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 408
Eyes | 42

6. Other Pre Specified Outcome: Cumulative Rates in Increased Intraocular Pressure (IOP) in All Eyes Attributed to Other Causes
Description: Rates of elevated intraocular pressure in all (primary + fellow) eyes attributed to other causes.
Time Frame: 1-6 hours postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | All Treated Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 408
Eyes | 0

7. Other Pre Specified Outcome: Cumulative Rates of Increased Intraocular Pressure (IOP) in All Eyes Attributed to Retained OVD
Description: as for outcome 5
Time Frame: Day 1 postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | All Treated Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 408
Eyes | 43

8. Other Pre Specified Outcome: Cumulative Rates of Increased Intraocular Pressure (IOP) in All Eyes Attributed to Other Causes
Description: Rates of elevated intraocular pressure in all (primary + fellow) eyes attributed to other causes.
Time Frame: Day 1 postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | All Treated Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 408
Eyes | 0

9. Other Pre Specified Outcome: Cumulative Rates of Increased Intraocular Pressure (IOP) in All Eyes Attributed to Retained OVD
Description: as for outcome 5
Time Frame: Day 5-9 postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | All Treated Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 408
Eyes | 43

10. Other Pre Specified Outcome: Cumulative Rates of Increased Intraocular Pressure (IOP) in All Eyes Attributed to Other Causes
Description: Rates of elevated intraocular pressure in all (primary + fellow) eyes attributed to other causes.
Time Frame: Day 5-9 postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | All Treated Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 408
Eyes | 1

11. Other Pre Specified Outcome: Cumulative Rates of Increased Intraocular Pressure (IOP) in All Eyes Attributed to Retained OVD
Description: as for outcome 5
Time Frame: Day 10-18 postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | All Treated Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 408
Eyes | 43

12. Other Pre Specified Outcome: Cumulative Rates of Increased Intraocular Pressure (IOP) in All Eyes Attributed to Other Causes
Description: Rates of elevated intraocular pressure in all (primary + fellow) eyes attributed to other causes
Time Frame: Day 10-18 postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | All Treated Eyes
Number analyzed (Participants) | 205
Number analyzed (Eyes) | 408
Eyes | 6

ADVERSE EVENTS:
Time Frame: Collection of adverse events began at the time of informed consent and continued until study completion (approximately 2-3 weeks)
Description: Serious Adverse Events (SAEs) (ocular and non-ocular) were collected. Non-serious non-ocular adverse events were not collected. The study protocol required that all secondary surgical interventions (SSIs) performed to treat an ocular SAE also be reported as SAEs.
Arm/Group | All Treated Eyes
All-Cause Mortality (participants affected / at risk) | 0/205
Serious Adverse Events (participants affected / at risk) | 2/408
Other Adverse Events (participants affected / at risk) | 45/408
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Eyes (N=408)
Incorrect EVO ICL Implantation (Eye disorders) | 1 (1)
Intraocular Lens Exchange (Eye disorders) | 1 (1)
Intraocular Cilium (Eye disorders) | 1 (1)
Surgery to Remove Intraocular Cilium (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Eyes (N=408)
Intraocular Pressure Increased (Eye disorders) | 45 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated from the study will be regarded as confidential, until appropriate analysis and review by the Sponsor or designee is completed. The results of the study may be published or presented by the Investigator(s) after review by, and in consultation and agreements with the Sponsor, and such that confidential or proprietary information is not disclosed. Prior to publication or presentation, a copy of the final text should be forwarded to the Sponsor or designee for comment.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT05538754/Prot_SAP_000.pdf